CLINICAL TRIAL: NCT06336928
Title: A Validation Study to Determine Concordance of Liquid Biopsy and Breast Cancer Diagnosis
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-23-6; NCI-2024-01332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-23-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma
Keywords: Liquid biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates whether a special type of blood analysis, called liquid biopsy (LBx), correlates with mammography results and/or diagnosis of breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the sensitivity of LBx for the presence of breast cancer in patient cohorts II. Determine the specificity of LBx for the presence of breast cancer in all patient cohorts.

OUTLINE: This is an observational study.

Patients undergo blood sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * Women

  * Age ≥ 18 years.
  * Screening Mammography Cohort: Patients who were referred for screening mammography and had mammography performed within 6 months prior to blood draw or will be undergoing mammography within 6 months after blood draw. Patient must not have personal history of breast cancer, history of breast biopsy or prior abnormal mammography findings are allowed. OR
  * Abnormal Screening Cohort: Patient who has had mammography that revealed abnormal results (BIRADS 3, 4, 5) or abnormal MRI results requiring further testing (additional imaging modality or biopsy). Patients must not have a history of breast cancer, history of breast biopsy, or prior abnormal mammography findings are allowed. The blood draw must occur in the time between the abnormal mammography and start of definitive treatment (surgery or neoadjuvant chemotherapy). Patients who have already undergone surgery/excisional biopsy due to abnormal mammography findings are not eligible. OR
  * New Beast Cancer Cohort: Patients with new biopsy proven diagnosis of breast cancer (invasive breast cancer or DCIS) within 60 days of blood draw who has not started any cancer directed therapy, including surgery, radiation, hormonal therapy or chemotherapy. Any breast cancer type patients at any stage are eligible. OR
  * Remission Breast Cancer Cohort: Patients with personal history of localized breast cancer (stage 1, 2, 3) that has been previously treated with cancer directed therapy, such as surgery, chemotherapy, radiation and/or hormonal therapy who has been in completed remission. Patients must complete their surgery, adjuvant chemotherapy and/or radiation therapy prior to enrollment. The blood draw must occur at least 90 days after completion of the specified treatment modalities. Patients on adjuvant hormonal therapy are eligible to enroll (those who are treated with adjuvant hormonal therapy in combination with CDK4/6 inhibitor must complete CDK4/6 inhibitor therapy prior to enrollment).

Exclusion Criteria:

* * Patients unable to give informed consent

  * Patients who have received blood transfusion with 14 days prior to study blood draw
  * Patients who had a heart attack, stroke, or pulmonary embolism within 3 months to study blood draw
  * Excisional breast biopsy in the prior 30 days. Needle biopsy of the breast is permitted

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referred for mammography, women newly diagnosed with breast cancer and completed no treatment, or women with history of localized breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2029-06-07 (Estimated); Study Completion 2030-06-07 (Estimated)

PRIMARY OUTCOMES:
Assess the sensitivity and specificity of LBx as a screening method for breast cancer | Up to 1 year
  LBx results using peripheral blood samples will be compared to a pathological diagnosis of breast cancer within 1 year of the liquid biopsy test.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Martynova, MD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California